CLINICAL TRIAL: NCT05011487
Title: Neoadjuvant Osimertinib Plus Chemotherapy for EGFR-mutant Stage III N2 Non-squamous Non-small Cell Lung Cancer
Brief Title: Neoadjuvant Osimertinib + Chemotherapy for EGFR-mutant Stage III NSCLC
Acronym: NOCE01
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yang Hong, Prof., Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SYSUCC B2021-167-01
Record Dates: First submitted 2021-08-15; First posted 2021-08-18 (Actual); Last update posted 2024-01-16 (Actual); Status verified 2024-01

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Non small cell lung cancer; neoadjuvant; EGFR-TKI
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — osimertinib; Cisplatin; Pemetrexed

STUDY DESIGN:
Intervention Model Description: osimertinib plus chemotherapy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- osimertinib plus chemotherapy (Experimental): Osimertinib (80mg/qd) po. for 60 days with two cycles of Pemetrexed (500 mg/m2) to be administered with cisplatin (75mg/m2) on Day 1 of every 3-week cycle for 2 cycles
  Interventions: Drug: Osimertinib; Drug: Cisplatin; Drug: Pemetrexed

INTERVENTIONS:
Drug: Osimertinib — 80mg/qd oral for 60 days
  Other Names: AZD9291; TAGRISSO
Drug: Cisplatin — Cisplatin (75mg/m2) to be administered with pemetrexed on Day 1 of every 3-week cycle for 2 cycles.
  Other Names: DDP
Drug: Pemetrexed — Pemetrexed (500 mg/m2) to be administered with cisplatin on Day 1 of every 3-week cycle for 2 cycles

SUMMARY:
This is a phase II, single-arm, multi-center study of neoadjuvant osimertinib in combination with chemotherapy for the treatment of patients with resectable EGFR-mutant stage III (N2) non-squamous non-small cell lung cancer

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically documented N2 positive non-squamous NSCLC with resectable (Stage IIIA or T3-4N2 IIIB) disease (according to Version 8 of the IASLC Cancer Staging Manual [IASLC Staging Manual in Thoracic Oncology 2016]).
* Complete surgical resection of the primary NSCLC must be deemed achievable, as assessed by a MDT evaluation (which should include a thoracic surgeon, specialized in oncologic procedures).
* Eastern Cooperative Oncology Group (ECOG) PS of 0 or 1 at enrolment, with no deterioration over the previous 2 weeks prior to baseline or day of first dosing
* A tumour which harbours one of the 2 common EGFR mutations known to be associated with EGFR-TKI sensitivity (Ex19del, L858R), either alone or in combination with other EGFR mutations (ie, T790M, G719X, Exon20 insertions, S7681 and L861Q).

Exclusion Criteria:

* Past medical history of ILD, drug-induced ILD, radiation pneumonitis which required steroid treatment, or any evidence of clinically active ILD.
* History of another primary malignancy, except for the following: Malignancy treated with curative intent and with no known active disease ≥2 years before the first dose of investigational product (IP) and of low potential risk for recurrence; Adequately treated non-melanoma skin cancer or lentigo malignancy without evidence of disease; Adequately treated carcinoma in situ without evidence of disease
* Patients who have pre-operative radiotherapy treatment as part of their care plan
* Mixed small cell and NSCLC histology
* T4 tumours infiltrating the aorta, the oesophagus and/or the heart; and/or any bulky N2 disease deemed unresectable
* Patients who are candidates to undergo only segmentectomies or wedge resections
* Prior treatment with any systemic anti-cancer therapy for NSCLC including chemotherapy, biologic therapy, immunotherapy, or any investigational drug
* Prior treatment with EGFR-TKI therapy
* Current use of (or unable to stop use prior to receiving the first dose of study treatment) medications or herbal supplements known to be strong inducers of cytochrome P450 (CYP) 3A4 (at least 3 weeks prior)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-08-13 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
complete lymph node clearance rate | From date of enrollment to an average of 12 weeks after the first dose
  the ratio of ypN0 percentage after resection

SECONDARY OUTCOMES:
Major Pathological Response (MPR) | From date of enrollment to an average of 12 weeks after the first dose
  Defined as ≤10% residual cancer cells in the main tumour, as assessed per central pathology laboratory post-surgery
Pathological complete response (pCR) | From date of enrollment to an average of 12 weeks after the first dose
  Defined as absence of any residual cancer cells in the dissected tumour samples, including the main tumour and lymph nodes, assessed post-surgery
Downstaging | From date of enrollment to an average of 12 weeks after the first dose
  Measured using pathologic mediastinal lymph node evaluation
Disease free survival (DFS) | From date of enrollment up to approximately 42 months after date of resection
  DFS is defined as the time from the date of surgery until the first date of disease recurrence (local or distant) or date of death due to any cause, whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: Hong Yang, Ph.D.,M.D., Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China